CLINICAL TRIAL: NCT05290935
Title: Anti-PD-1 Antibody Camrelizumab Combined With Albumin-bound Paclitaxel for Recurrent and Persistent Advanced Cervical Cancer Refractory to Platinum-based Chemotherapy: A Single Arm, Multi-Center, Open, Phase II Trial
Brief Title: Immunotherapy for Recurrent Cervical Cancer Refractory to Platinum-based Chemotherapy: Multi-Center Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REPACC-3
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Cervical Carcinoma; Persistent Advanced Cervical Carcinoma; Chemotherapy; Immune Checkpoint Inhibitors; Anti-PD-1 Antibody; Albumin-bound Paclitaxel
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): The patients in the study group would accept the treatment of a combination of anti-PD-1 antibody camrelizumab and albumin-bound paclitaxel.
  Interventions: Drug: Anti-PD-1 antibody camrelizumab; Drug: Albumin-bound paclitaxel

INTERVENTIONS:
Drug: Anti-PD-1 antibody camrelizumab — Camrelizumab: 200 mg every time, every 3 weeks, which would be sustained until the appearance of disease progression on intolerable adverse events, and no more than 24 months
Drug: Albumin-bound paclitaxel — Albumin-bound paclitaxel: 200-300 mg every time, every 3 weeks, no more than 6 courses

SUMMARY:
This is a updated trial of NCT04188860 as a multi-center study. For recurrent or persistent advanced cervical cancer patients, the first-line chemotherapy was based on platinum. However, if they were refractory to platinum-based chemotherapy, there were no other more effective medications or treatment. The marketing of anti-PD-1 antibody has provided an opportunity of curative management. This single arm, open, phase II trial would recruit 122 eligible patients. A combination of anti-PD-1 antibody camrelizumab and albumin-bound paclitaxel would be given for all patients. The primary end is overall response rate (ORR). The second ends include progression-free survival, overall survival, disease control rate, remission duration, and adverse events. A molecular testing, mainly consisting of genomic analysis, will be carried in the oncologic tissues.

ELIGIBILITY:
Inclusion Criteria:

* Female of 18-75 years old
* Eastern Cooperative Oncology Group score 0-1
* Pathological confirmed of uterine cervical adenocarcinoma, squamous carcinoma, or adenosquamous carcinoma, with stage IA1 (with lymph-vascular space invasion) to IVB, which had accepted radical treatment for the purpose of cure
* Having accepted at least one regimen of platinum-based chemotherapy after the diagnosis of recurrent or persistent advanced cervical cancer, and having an interval of at least 4 weeks since fulfilling the last treatment regimen
* At least one measurable lesion defined by Response Evaluation Criteria in Solid Tumors (RECIST) guideline 1.1
* Anticipative survival period of 3 months or more
* Lab testing within reference ranges
* With appropriate contraception
* Provided consents of participating the trial

Exclusion Criteria:

* With brain metastasis
* With addiction to psychiatric medications or with mental disorders
* With following history and/or complications: autoimmune disease; systematic utilization of corticosteroids (with equivalent of prednison of > 10 mg/day) or other immunosuppressors within 14 days; utilization of antitumor vaccine or other immunostimulation treatment with 3 months; exposure to PD-1 antibody, or PD-L1 antibody, or PD-L2 antibody, or cytotoxic T lymphocyte-associated antigen-4 antibody; history of other malignancies; pulmonary tuberculosis; interstitial pneumonia or related history; active hepatitis; positive testing of human immunodeficiency
* With adverse effects more than Common Terminology Criteria for Adverse Events grade 1 (except for alopecia), which caused by previous anti-tumor treatment
* With infective disease which need systematic treatment within 14 days
* With severe open trauma, fracture or major surgery with past 4 weeks
* With potential allergy or intolerance to study regimens
* Not eligible for the study judged by researchers

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-03-13 (Actual); Primary Completion 2022-12-13 (Estimated); Study Completion 2024-03-13 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | One year
  The rates of complete and partial remission

SECONDARY OUTCOMES:
Progression-free survival | One year
  The length of time during and after the treatment of the cancer, that a patient lives with the disease but it does not get worse
Overall survival | One year
  The length of time from either the date of diagnosis or the start of treatment for the cancer, that patients diagnosed with the disease are still alive
Disease control rate | One year
  The rates of complete and partial remission, and stable disease
Adverse event rates | One year
  The rates of adverse events judged by Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China